CLINICAL TRIAL: NCT01065480
Title: Training Motivational Interviewing Using Live Supervision
Brief Title: Training Clinicians in Motivational Interviewing
Acronym: MITraining
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Edward Nunes, Professor of Clinical Psychiatry, New York State Psychiatric Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: #6052/7087R; R01DA016950 (NIH)
Record Dates: First submitted 2010-02-08; First posted 2010-02-09 (Estimated); Results first posted 2017-11-06 (Actual); Last update posted 2018-12-26 (Actual); Status verified 2018-12

CONDITIONS: Substance Abuse
Keywords: Training; Substance Abuse; Counseling; Motivational Interviewing
MeSH Terms: conditions — Substance-Related Disorders | interventions — Motivational Interviewing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Live Teleconference Supervision (Active Comparator): Clinicians from participating substance abuse treatment programs receive live supervision by MI trainer via teleconference while in session with client.
  Interventions: Behavioral: Live teleconference supervision
- Taped Review Supervision (Active Comparator): Clinicians from participating substance treatment programs audio record session with client and receive supervision after the session by MI trainer.
  Interventions: Behavioral: Taped Review Supervision

INTERVENTIONS:
Behavioral: Live teleconference supervision — Participants receive live teleconference supervision during a session with a client on their use of Motivational Interviewing (MI) in the session. MI is a directive, client-centered counseling style for eliciting behavior change by helping clients to explore and resolve ambivalence. Compared with nondirective counselling, it is more focused and goal-directed. The examination and resolution of ambivalence is its central purpose, and the counselor is intentionally directive in pursuing this goal.
  Other Names: Motivational Enhancement Therapy; MI; MET
  Arms: Live Teleconference Supervision
Behavioral: Taped Review Supervision — Participants audio record a session with a client and receive supervision after the session on their use of Motivational Interviewing during the session.
  Arms: Taped Review Supervision

SUMMARY:
This study aims to train Substance Abuse Treatment Clinicians in the use of Motivational Interviewing techniques through live supervision.

DETAILED DESCRIPTION:
New evidence-based treatments have been slow to be adopted into the routine practice of addiction treatment, and traditional training methods are of limited effectiveness. In this study, the investigators propose to continue development of methods for training clinicians in Motivational Interviewing (MI), based on the principle of live supervision. Live supervision (supervisor and trainee seeing a patient together) is common in basic training, but rarely used in continuing education. In the initial funding period we developed Teleconference Supervision (TCS), which implements live supervision by an expert through teleconferencing technology, harnessing the principles of context-dependent learning, differential reinforcement with immediacy of feedback, and modeling. Clinicians interview standard patients at their home clinics, while Supervisors listen via telephone. The clinician wears an earpiece, through which the Supervisor provides immediate feedback and coaching designed to differentially reinforce and shape MI skills. In a randomized controlled trial with community clinicians (N= 100), TCS produced superior overall MI skill, compared to control conditions where clinicians received Workshop only training, or standard tape-based supervision. Findings were encouraging yet the proportion of clinicians achieving expert proficiency was limited, and there were trends toward loss of skill at follow-up, suggesting longer training is needed to maximize and sustain MI skill.

In the new funding period, the investigators propose to build and improve upon TCS by testing an extended model of Teleconference Supervision (TCS-Plus), which will preserve the elements of live supervision from an expert supervisor but will also provide 4 sessions of enhanced tape review supervision on a bi-weekly basis after the initial TCS training. Using telephone technology, enhanced taped review allows the Supervisor and Clinician to listen to the taped session together before discussing the session. Practice sessions will increase from 5 to 9 and be spread out from 8 to 16 weeks. Providing both TCS and enhanced tape review supervision maximizes supervision style advantages. While both offer context dependent learning, TCS provides for modeling and differential reinforcement with immediacy of feedback, and enhanced tape review provides ample time to role play and discuss technique. TCS-Plus will be compared to standard Tape Review supervision. The proposed project will be a StageI trial, intent on maximizing the gains already detected with the TCS model. The investiators will assess if TCS-Plus produces superior MI skill to standard Tape Review supervision in a randomized trial with 130 community based-clinicians. It is hoped that, if successful, TCS-Plus could be a model for remote training and supervision at community treatment programs, promoting adoption of a variety of evidence-based treatments for substance use disorders into routine practice.

ELIGIBILITY:
Inclusion Criteria:

1. Clinician, aged 18 to 75, employed in good standing at least 50% time at a licensed substance abuse treatment program.
2. Carries a regular caseload of patients or clients for whom he/she serves as primary therapist.
3. Interested in learning Motivational Interviewing and willing to follow treatment guidelines and training protocol, including random assignment to groups.
4. Willing and able to attend a 2 day workshop, to tape subsequent sessions with patients for evaluation of MI skillfulness by Training Team members and raters, and to participate in supervision, including taping of sessions for review by Training Team members and raters and/or having supervisor listen to, and comment on, live sessions.

Exclusion Criteria:

1. Planning to terminate employment at the current treatment program within the next six months.
2. Has received credentialing as a Motivational Interviewing trainer, or served as a Motivational Interviewing or Motivational Enhancement Therapy therapist in a clinical trial which provided feedback on MI skill.
3. Has received formal training in Motivational Interviewing within the last three months

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2010-03-01 (Actual); Primary Completion 2015-06-01 (Actual); Study Completion 2015-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edward V Nunes, MD, Principal Investigator — New York State Psychiatric Institute/Columbia University
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Live Teleconference Supervision | Taped Review Supervision
Started | 48 | 43
Completed | 48 | 43
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Live Teleconference Supervision | Taped Review Supervision | Total
Number analyzed (Participants) | 48 | 43 | 91
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 48 | 43 | 91
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 20 | 49
  Male | 19 | 23 | 42
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: White, not Hispanic | 12 | 11 | 23
  Race/Ethnicity: Black, not Hispanic | 24 | 14 | 38
  Race/Ethnicity: Hispanic | 12 | 15 | 27
  Race/Ethnicity: Asian or Pacific Islander | 0 | 2 | 2
  Race/Ethnicity: American Indian or Native American | 0 | 0 | 0
  Race/Ethnicity: Other | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 48 | 43 | 91

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With MI Skillfulness
Description: MI skillfulness measured by the Motivational Interviewing Treatment Integrity Scale (MITI) on double coded audio recorded sessions and clinical interviews. The cumulative number of participants with MI Skillfulness at each time point assessed at 1, 8, 16, 24, and 32 weeks are reported.
Time Frame: 1,8,16, 24 and 32 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Live Teleconference Supervision | Taped Review Supervision
Number analyzed (Participants) | 48 | 43
Participants | 48 | 43

ADVERSE EVENTS:
Time Frame: From consent through completion of trial, an average of 4 weeks.
Arm/Group | Live Teleconference Supervision | Taped Review Supervision
All-Cause Mortality (participants affected / at risk) | 0/48 | 0/43
Serious Adverse Events (participants affected / at risk) | 0/48 | 0/43
Other Adverse Events (participants affected / at risk) | 0/48 | 0/43

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No